CLINICAL TRIAL: NCT05528861
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Lirentelimab in Adult Subjects With H-1 Antihistamine Refractory Chronic Spontaneous Urticaria
Brief Title: A Study to Assess Subcutaneous Lirentelimab (AK002) in Chronic Spontaneous Urticaria
Acronym: MAVERICK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No longer pursuing development
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK002-027
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Chronic Spontaneous Urticaria; Chronic Urticaria; Urticaria; Chronic Idiopathic Urticaria; Chronic Autoimmune Urticaria; Idiopathic Chronic Urticaria; Autoimmune Urticaria
MeSH Terms: conditions — Chronic Urticaria; Urticaria | interventions — AK002

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lirentelimab (AK002) (Experimental): Subjects in this arm will receive lirentelimab (AK002) administered subcutaneously.
  Interventions: Drug: Lirentelimab (AK002)
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lirentelimab (AK002) — Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8
  Other Names: AK002
  Arms: Lirentelimab (AK002)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of subcutaneous lirentelimab (AK002) in adult subjects with H-1 antihistamine refractory chronic spontaneous urticaria. Subjects who complete the randomized, double-blind, placebo-controlled treatment period may have the option to enroll in an open-label extension period and receive up to 6 doses of subcutaneous lirentelimab.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject is able to understand the information on the study, has the capacity to consent, and has provided written informed consent.
2. Male and female subjects ≥18 years of age at the time of screening.
3. CSU diagnosis for ≥6 months.
4. Diagnosis of moderate-severe CSU refractory to H1-antihistamine (H1-AH) at a minimum of the licensed dose at the licensed frequency at the time of randomization as defined by the following: presence of hives and itch for ≥6 consecutive weeks prior to Screening Visit 1; UAS7 score (range 0-42) ≥16 and HSS7 score (range 0-21) ≥8 during the 7 days prior to randomization.
5. Subjects that are omalizumab-naïve or omalizumab-exposed.
6. Subjects must be on stable dose of H1-AH, between 1x and 4x of the licensed dose and at the licensed frequency, for treatment of CSU for at least 1 week prior to screening and willing to remain on a stable dose throughout the study.
7. Able and compliant with completing a daily symptom eDiary for the duration of the study and adherent to the study visit schedules.

Key Exclusion Criteria:

1. History of hypersensitivity to the study drugs or their excipients or to drugs of similar chemical classes (i.e., murine, chimeric or human antibodies).
2. Current use of biologics for any indication.
3. Demonstrated lack of primary response to treatment with a biologic therapy (e.g., omalizumab) for the treatment of CSU.
4. Use of any of the following treatments within 4 weeks prior to the baseline visit or any condition that in the opinion of the Investigator is likely to require such treatment(s) during the first 4 weeks of study treatment: (i) immunosuppressive or immunomodulatory drugs, including but not limited to systemic calcineurin inhibitors (e.g., cyclosporin, tacrolimus), mTOR inhibitors (e.g., sirolimus, everolimus), anti-metabolites (e.g., azathioprine, methotrexate, 6-mercaptopurine, leflunomide, mycophenolate mofetil), alkylating agents (e.g., cyclophosphamide), TNF inhibitors (e.g., infliximab, adalimumab), and eosinophil-depleting drugs (e.g., benralizumab, pramipexole); (ii) routine (daily or every other day during 5 or more consecutive days) doses of systemic hydroxychloroquine; (iii) intravenous immunoglobulin (IVIG); (iv) plasmapheresis.
5. Use of oral Janus kinase (JAK) inhibitors within 8 weeks of the baseline visit.
6. Use of any of the following treatments within 3 weeks prior to the baseline visit: (i) H2 antihistamines (H2-AH); (ii) routine (daily or every other day during 5 or more consecutive days) doses of systemic corticosteroids; (iii) regular (daily or every other day) doxepin (oral); (iv) leukotriene receptor antagonists (LTRA) (e.g., montelukast, zafirlukast).
7. H1-AH use at greater than approved doses or greater than local CSU guideline recommended doses after Screening Visit 1.
8. Previous treatment with biologics: (i) any cell-depleting agents including but not limited to rituximab within 6 months prior to the baseline visit or until lymphocyte count returns to normal, whichever is longer; (ii) other biologics, including investigational biologics (e.g., dupilumab, omalizumab, benralizumab, etc) within 5 half-lives if known or 8 weeks prior to the baseline visit, whichever is longer.
9. Planned or anticipated use of any prohibited medication.
10. Subjects having causes other than CSU for their urticaria including symptomatic dermographism, cholinergic urticaria, or any inducible urticaria.
11. Subjects with known or suspected urticarial vasculitis.
12. Subjects with known or suspected hereditary angioedema.
13. Any other skin disease associated with chronic itch, including atopic dermatitis, that in the Investigator's opinion might influence study outcome and subject's interpretation of symptoms caused by CSU.
14. A helminth parasitic infection diagnosed within 6 months prior to the date that informed consent is obtained and has not been treated with or has failed to respond to standard-of-care therapy.
15. Participation in a concurrent interventional study with the last intervention occurring within 30 days prior to study drug administration (or 90 days or 5 half-lives, whichever is longer, for biologic products).
16. Vaccination with live attenuated vaccines within 30 days prior to initiation of treatment in the study, during the treatment period, or vaccination expected within 5 half-lives (4 months) of study drug administration. This exclusion criterion does not apply to all types and formulations of vaccines (including live attenuated vaccines) currently authorized/approved by FDA or other regulatory authority for the prevention of COVID-19, which may be administered before, during, or after the study. The vaccine should not be administered within 3 days before and within 3 days after the administration of lirentelimab so that any side effects caused by either of the 2 medications can more easily be determined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chin Lee, MD, MPH, Study Director — Allakos Inc.
Locations (67):
- United States (51):
  - Allakos Investigational Site 227-024, Birmingham, Alabama
  - Allakos Investigational Site 227-068, Cullman, Alabama
  - Allakos Investigational Site 227-014, Phoenix, Arizona
  - Allakos Investigational Site 227-023, Scottsdale, Arizona
  - Allakos Investigational Site 227-058, Bakersfield, California
  - Allakos Investigational Site 227-026, Los Angeles, California
  - Allakos Investigational Site 227-009, Los Angeles, California
  - Allakos Investigational Site 227-011, Mission Viejo, California
  - Allakos Investigational Site 227-021, Santa Monica, California
  - Allakos Investigational Site 227-031, Upland, California
  - Allakos Investigational Site 227-006, Colorado Springs, Colorado
  - Allakos Investigational Site 227-036, Jacksonville, Florida
  - Allakos Investigational Site 227-062, Miami, Florida
  - Allakos Investigational Site 227-041, Sarasota, Florida
  - Allakos Investigational Site 227-067, Tampa, Florida
  - Allakos Investigational Site 227-005, Tampa, Florida
  - Allakos Investigational Site 227-018, Columbus, Georgia
  - Allakos Investigational Site 227-045, Boise, Idaho
  - Allakos Investigational Site 227-045, Normal, Illinois
  - Allakos Investigational Site 227-057, River Forest, Illinois
  - Allakos Investigational Site 227-074, Plainfield, Indiana
  - Allakos Investigational Site 227-047, Overland Park, Kansas
  - Allakos Investigational Site 227-051, Lexington, Kentucky
  - Allakos Investigational Site 227-019, Baltimore, Maryland
  - Allakos Investigational Site 227-012, Towson, Maryland
  - Allakos Investigational Site 227-063, White Marsh, Maryland
  - Allakos Investigational Site 227-016, Boston, Massachusetts
  - Allakos Investigational Site 227-034, Ann Arbor, Michigan
  - Allakos Investigational Site 227-032, Detroit, Michigan
  - Allakos Investigational Site 227-070, Farmington Hills, Michigan
  - Allakos Investigational Site 227-073, Dilworth, Minnesota
  - Allakos Investigational Site 227-052, Rochester, Minnesota
  - Allakos Investigational Site 227-008, St Louis, Missouri
  - Allakos Investigational Site 227-059, Missoula, Montana
  - Allakos Investigational Site 227-022, Brooklyn, New York
  - Allakos Investigational Site 227-007, Great Neck, New York
  - Allakos Investigational Site 227-002, Asheville, North Carolina
  - Allakos Investigational Site 227-013, Cincinnati, Ohio
  - Allakos Investigational Site 227-029, Cincinnati, Ohio
  - Allakos Investigational Site 227-043, Columbus, Ohio
  - Allakos Investigational Site 227-064, Toledo, Ohio
  - Allakos Investigational Site 227-060, Oklahoma City, Oklahoma
  - Allakos Investigational Site 227-027, Portland, Oregon
  - Allakos Investigational Site 227-028, Hershey, Pennsylvania
  - Allakos Investigational Site 227-040, Philadelphia, Pennsylvania
  - Allakos Investigational Site 227-066, North Charleston, South Carolina
  - Allakos Investigational Site 227-055, Austin, Texas
  - Allakos Investigational Site 227-049, El Paso, Texas
  - Allakos Investigational Site 227-039, Murray, Utah
  - Allakos Investigational Site 227-071, Murray, Utah
  - Allakos Investigational Site 227-033, Greenfield, Wisconsin
- Germany (12):
  - Allakos Investigational Site 227-204, Augsburg
  - Allakos Investigational Site 227-201, Berlin
  - Allakos Investigational Site 227-214, Buxtehude
  - Allakos Investigational Site 227-205, Darmstadt
  - Allakos Investigational Site 227-209, Erlangen
  - Allakos Investigational Site 227-208, Frankfurt
  - Allakos Investigational Site 227-207, Langenau
  - Allakos Investigational Site 227-203, Leipzig
  - Allakos Investigational Site 227-210, Mainz
  - Allakos Investigational Site 227-202, Mainz
  - Allakos Investigational Site 227-211, Munich
  - Allakos Investigational Site 227-206, Osnabrück
- Poland (4):
  - Allakos Investigational Site 227-302, Lodz
  - Allakos Investigational Site 227-304, Lodz
  - Allakos Investigational Site 227-303, Lublin
  - Allakos Investigational Site 227-301, Zabrze

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 127 subjects who were enrolled in the main study received up to 6 doses of AK002 or placebo. 117 subjects from the main study continued into the open-label extension (OLE) period and received up to 6 doses of AK002.
Groups:
- AK002 SC 300 mg (Main Study) - AK002 Continuing (OLE): For the main study period, subjects in this arm received up to 6 doses of 300 mg of lirentelimab (AK002) administered subcutaneously (SC) every 2 weeks.
  For the open-label extension (OLE) period, subjects who completed the main study and met eligibility criteria had the option to receive up to 6 doses of AK002 SC.
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8
- Placebo (Main Study) - Placebo Rollover (OLE): For the main study period, subjects in this arm received up to 6 doses of placebo administered subcutaneously every 2 weeks.
  For the open-label extension (OLE) period, subjects who completed the main study and met eligibility criteria had the option to rollover and receive up to 6 doses of 300 mg AK002 SC.
  Placebo: Placebo
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8
Period: Main Study
Arm/Group | AK002 SC 300 mg (Main Study) - AK002 Continuing (OLE) | Placebo (Main Study) - Placebo Rollover (OLE)
Started | 66 | 61
Completed | 60 | 57
Not Completed | 6 | 4
Period: Open-Label Extension
Arm/Group | AK002 SC 300 mg (Main Study) - AK002 Continuing (OLE) | Placebo (Main Study) - Placebo Rollover (OLE)
Started | 60 | 57
Completed | 27 | 30
Not Completed | 33 | 27

BASELINE CHARACTERISTICS:
Population: Baseline analysis is reported on the safety population of the main study period. Baseline information of OLE subjects is not reported since it is already captured as part of the main study population.
Groups:
- AK002 SC 300 mg (Main Study): Subjects in this arm received up to 6 doses of 300 mg of lirentelimab (AK002) administered subcutaneously every 2 weeks in the main study.
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8
- Placebo (Main Study): Subjects in this arm received up to 6 doses of placebo administered subcutaneously every 2 weeks in the main study.
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study) | Total
Number analyzed (Participants) | 66 | 61 | 127
Age, Continuous [Median (Full Range); unit: years] | 41 [19 to 77] | 43 [24 to 76] | 41 [19 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 57 | 107
  Male | 16 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 56 | 51 | 107
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 54 | 43 | 97
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 55 | 112
  Poland | 2 | 1 | 3
  Germany | 7 | 5 | 12
Weekly Urticaria Assessment Score (UAS7) [Mean (Standard Deviation); unit: Score on a scale] — The UAS7 is the sum for 7 days of the daily Hives Severity Score (HSS) and the daily Itch Severity Score (ISS). The daily HSS is recorded on a scale of 0 (none) to 3 (>50 hives) and the daily ISS is recorded on a scale of 0 (none) to 3 (severe). Therefore, the possible range of the weekly UAS7 score is 0-42, with 42 being the most severe.
  Score on a scale | 31.0 (7.4) | 31.9 (7.8) | 31.4 (7.6)
Weekly Hive Severity Score (HSS7) [Mean (Standard Deviation); unit: Score on a scale] — The severity of hives will be recorded on a scale of 0 (none) to 3 (> 50 hives). A weekly Hives Severity score (HSS7) is derived by adding the average daily scores of the 7 days preceding the visit. Therefore, the possible range of the weekly score is 0 - 21.
  Score on a scale | 14.9 (4.2) | 15.8 (4.0) | 15.3 (4.2)
Weekly Itch Severity Score (ISS7) [Mean (Standard Deviation); unit: Score on a scale] — The severity of itching will be recorded on a scale of 0 (none) to 3 (severe). A weekly Itch Severity Score (ISS7) is derived by adding the average daily scores of the 7 days preceding the visit. Therefore, the possible range of the weekly score is 0 - 21.
  Score on a scale | 16.1 (4.4) | 16.1 (4.3) | 16.1 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Weekly Urticaria Assessment Score (UAS7) From Baseline at Week 12
Description: The UAS7 is the sum for 7 days of the daily Hives Severity Score (HSS) and the daily Itch Severity Score (ISS). The daily HSS is recorded on a scale of 0 (none) to 3 (>50 hives) and the daily ISS is recorded on a scale of 0 (none) to 3 (severe). Therefore, the possible range of the weekly UAS7 score is 0-42, with 42 being the most severe.
Time Frame: Baseline to Week 12
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 64 | 59
score on a scale | -7.9 (1.9) | -8.4 (2.0)
Statistical Analysis 1: Comparison: AK002 SC 300 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.8174, ANCOVA; LSM Difference from Placebo = 0.5, 95% CI 2-sided [-3.6 to 4.5], Standard Error of Mean 2.1

2. Secondary Outcome: Absolute Change in Hives Severity Score (HSS7) From Baseline at Week 12
Description: The severity of hives will be recorded by all subjects once daily on a scale of 0 (none) to 3 (> 50 hives). A weekly HSS score (HSS7) is derived by adding the average daily scores of the 7 days preceding the visit. Therefore, the possible range of the weekly score is 0 - 21.
Time Frame: Baseline to Week 12
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 64 | 59
score on a scale | -4.0 (0.8) | -4.6 (0.9)
Statistical Analysis 1: Comparison: AK002 SC 300 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.5857, Mixed Models Analysis; LSM Difference from Placebo = 0.6, 95% CI 2-sided [-1.6 to 2.8], Standard Error of Mean 1.1

3. Secondary Outcome: Absolute Change in Itch Severity Score (ISS7) From Baseline at Week 12
Description: The severity of itching will be recorded by all subjects once daily on a scale of 0 (none) to 3 (severe). A weekly ISS score (ISS7) is derived by adding the average daily scores of the 7 days preceding the visit. Therefore, the possible range of the weekly score is 0 - 21.
Time Frame: Baseline to Week 12
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 64 | 59
score on a scale | -4.4 (0.8) | -4.3 (0.9)
Statistical Analysis 1: Comparison: AK002 SC 300 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.9633, Mixed Models Analysis; LSM Difference from Placebo = -0.1, 95% CI 2-sided [-2.2 to 2.1], Standard Error of Mean 1.1

4. Secondary Outcome: Proportion of Subjects Achieving Weekly Urticaria Assessment Score (UAS7)=0 at Week 12
Description: The UAS7 is the sum for 7 days of the daily Hives Severity Score (HSS) and the daily Itch Severity Score (ISS). The possible range of the UAS7 is 0-42.
Time Frame: At Week 12
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 64 | 59
percentage of participants | 6.3 | 0
Statistical Analysis 1: Comparison: AK002 SC 300 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.1201, Fisher Exact; Risk Difference (RD) = 6.25, 95% CI 2-sided [-11.40 to 23.78]

5. Other Pre Specified Outcome: Safety and Tolerability of up to 6 Doses of Open-label AK002 in Subjects With Chronic Spontaneous Urticaria in the Open-label Extension Period
Description: Adverse events were assessed throughout the open-label extension period.
Time Frame: Through study completion, up to 34 weeks (open-label extension period)
Measure: Count of Participants; unit: Participants
Groups:
- AK002 Continuing (OLE): Subjects in this arm received AK002 in the main study and continued to receive up to 6 doses of 300 mg AK002 SC in the open-label extension (OLE) period.
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1(IgG1)monoclonal antibody directed against Siglec-8
- Placebo Rollover (OLE): Subjects in this arm received placebo in the main study and rolled over to receive up to 6 doses of 300 mg AK002 SC in the open-label extension (OLE) period.
  Placebo: Placebo AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1(IgG1)monoclonal antibody directed against Siglec-8
Arm/Group | AK002 Continuing (OLE) | Placebo Rollover (OLE)
Number analyzed (Participants) | 60 | 57
Participants
  Subjects with ≥1 adverse events | 31 | 26
  Subjects with ≥1 treatment-related adverse events | 6 | 12
  Subjects with an adverse event leading to study drug discontinuation | 4 | 1
  Subjects with ≥1 serious adverse events | 2 | 2
  Subjects with ≥1 treatment-related serious adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, up to 34 weeks (open-label extension period)
Groups:
- AK002 Continuing (OLE): Subjects in this arm received AK002 in the main study and continued to receive up to 6 doses of 300 mg AK002 SC in the open-label extension (OLE) period.
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8
- Placebo Rollover (OLE): Subjects in this arm received placebo in the main study and rolled over to receive up to 6 doses of 300 mg AK002 SC in the open-label extension (OLE) period.
  Placebo: Placebo
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study) | AK002 Continuing (OLE) | Placebo Rollover (OLE)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/61 | 0/60 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/66 | 1/61 | 2/60 | 2/57
Other Adverse Events (participants affected / at risk) | 26/66 | 18/61 | 22/60 | 19/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AK002 SC 300 mg (Main Study) (N=66) | Placebo (Main Study) (N=61) | AK002 Continuing (OLE) (N=60) | Placebo Rollover (OLE) (N=57)
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
Epiglottitis obstructive (Infections and infestations) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AK002 SC 300 mg (Main Study) (N=66) | Placebo (Main Study) (N=61) | AK002 Continuing (OLE) (N=60) | Placebo Rollover (OLE) (N=57)
Injection site reaction (General disorders) | 14 | 6 | 4 | 9
Nasopharyngitis (Infections and infestations) | 6 | 3 | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 3 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 12 | 5 | 1 | 5
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 2 | 3 | 6 | 2
Urinary tract infection (Infections and infestations) | 2 | 3 | 5 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 3 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement contains a limit on publication of results following completion of the trial. PIs are not allowed to publish results until a joint publication for the multicenter study or a set period of time. After that time, PIs may only publish results from their portion of the study.

DOCUMENTS (2):
  • Study Protocol (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT05528861/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT05528861/SAP_001.pdf